CLINICAL TRIAL: NCT04848571
Title: Effects of Chinese Medicine on Early Pregnant Women
Status: Completed | Type: Observational
Sponsor: Shanghai Meiji Health Science and Technology Co., Ltd. (Industry)
Collaborators: Shanghai Institute of Palnned parenthood research (Unknown)
Responsible Party: Sponsor
Other Study IDs: sippr
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pregnant Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Pregnant women who received IVF and not taken Chinesene fetal protection medicine until sampling
- medicine group: Pregnant women who received IVF and have taken Chinesene fetal protection medicine from the fourth week during early pregnancy
  Interventions: Combination Product: Fetal Protection Pill

INTERVENTIONS:
Combination Product: Fetal Protection Pill — A Chinese medicine used in pregnant women for fetal protection, including mainly Rehmannia glutinosa.
  Groups: medicine group

SUMMARY:
From April 2021 to December 2021, 45 pregnant women who received intro fertilization-embyro transfer (IVF-ET) were recuited. According to their own wishes, 28 of them took Chinese medicine from the 2nd week after embryo transfer (intervention group), while the remaining 17 did not intake Chinese medicine (control group). Blood and feces samples were collected in the early morning of the 4th week after embryo transfer to detect 16S DNA sequences in feces, plasma metabolites, and whole blood transcriptomics.

DETAILED DESCRIPTION:
Investigators planned to performed a observational clinical trial to determine the effects of the Chinese medicine (Gushen Antai recipe) including mainly Rehmannia glutinosa used in pregnant women for fetal protection. Two groupswere recruited, Chinese medicine intervention group and control group without Chinese medicine. In the 4th week after embryo transfer, blood and fetal were sampled for metabolic and intestinal microbiota analysis.

ELIGIBILITY:
Inclusion Criteria:

* recieved IVF
* childbirth without miscarriage
* taking vitamins during pregnancy

Exclusion Criteria:

* miscarrige
* missed sampling in the fourth week of pregnancy
* not appropriate judged by the doctor

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: 17 patients in contol group and 28 patients in the Chinaese medicine intervention group
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
16s DNA analysis in feces | the fourth week in early pregnancy
  intestinal flora analysis in patients

SECONDARY OUTCOMES:
plasma metabonomics analysis by GC/LC mass | the fourth week in early pregnancy
  plasma metabolic analysis in patients

OTHER OUTCOMES:
whole blood transcriptomics analysis by RNA sequencing | the fourth week in early pregnancy
  blood transcriptomic analysis in patients

CONTACTS AND LOCATIONS:
Overall Officials: Enuo Liu, Dr., Study Chair — Shanghai Institute of Planned Parenthood Research
Locations (1):
- Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No